CLINICAL TRIAL: NCT06369038
Title: Assessment of Dental Anxiety After Children's Drawing as a Projective Tool During Dental Extraction Under Local Anesthesia - A Diagnostic Accuracy Test Study.
Brief Title: Children's Drawing as a Projective Tool to Assess Dental Anxiety
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Weam Sayed Abd El Mautie, pediatric dental resident at faculty of dentistry Cairo university, Cairo University
Other Study IDs: CUP3222024
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; drawing; projective tool

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: observation of level of dental anxiety in children — analysis of children's drawings using CD:H index

SUMMARY:
The aim in this study is to compare the results of anxiety measurement of the child using the CD:H scale with the long-used Face,Legs,Activity,Cry and Consolability scale (FLACC scale) , Frankl behaviour rating scale and pulse oximeter reading, to see if the drawing alone can be a reliable tool to predict the child's behaviour before the dental procedure.

DETAILED DESCRIPTION:
Dental anxiety is one of the major problems facing us in pediatric dentistry, the new experience that the child has to go through together with the difficulty for the child to express his exact cause of fear increases the problem.

Research has shown that healthcare providers spend more time communicating with parents than pediatric patients. In a typical medical care visit, less than 20% of the communication engaged pediatric patients, regardless of age. Most decision-making and treatment planning are done by dentists and parents.

Even when the dentist tries to engage the child in the conversation it usually includes the social aspect "his favourite hobby, toys, school topics, etc…" rather than the medical history or treatment decisions so the child is unaccustomed to discussing his dental fears and complaints to the dentist, hence we lose a lot of the child's trust.

Drawing has been used in literature as a psychological method to express one's thoughts and fears and can be analyzed by the healthcare provider to know the deeper thoughts of the child.

Thus, the current study aims to deeply understand the children's point of view towards dental treatment and use the drawings as a projective tool to assess the dental anxiety in those children by simple index and defined scores that every dentist could learn and apply.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 6 to 12 years.
* Children with past dental experience.
* One or more primary teeth indicated for simple extraction procedure.

Exclusion Criteria:

* Patients lacking cooperative behavior (very young age and patients with certain medical or psychological disorders) according to Wright's classification.
* Refusal of participation.
* Lack of informed consent by the child's parents.
* If the child shows any signs of disinterest in drawing.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with previous dental experience aging from 6 to 12 years and have one or more teeth indicated for simple extraction.
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
FLAAC behavioral scale | 6 months
  scale to measure the level of anxiety for children during dental visit

CONTACTS AND LOCATIONS:
Overall Officials: Weam S Ayoub, MsC, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cianetti S, Lombardo G, Lupatelli E, Pagano S, Abraha I, Montedori A, Caruso S, Gatto R, De Giorgio S, Salvato R. Dental fear/anxiety among children and adolescents. A systematic review. Eur J Paediatr Dent. 2017 Jun;18(2):121-130. doi: 10.23804/ejpd.2017.18.02.07. PMID 28598183
- [Background] Facco E, Zanette G, Favero L, Bacci C, Sivolella S, Cavallin F, Manani G. Toward the validation of visual analogue scale for anxiety. Anesth Prog. 2011 Spring;58(1):8-13. doi: 10.2344/0003-3006-58.1.8. PMID 21410359
- [Background] Clatworthy S, Simon K, Tiedeman ME. Child drawing: hospital--an instrument designed to measure the emotional status of hospitalized school-aged children. J Pediatr Nurs. 1999 Feb;14(1):2-9. doi: 10.1016/S0882-5963(99)80054-2. PMID 10063243
- [Background] Voepel-Lewis T, Zanotti J, Dammeyer JA, Merkel S. Reliability and validity of the face, legs, activity, cry, consolability behavioral tool in assessing acute pain in critically ill patients. Am J Crit Care. 2010 Jan;19(1):55-61; quiz 62. doi: 10.4037/ajcc2010624. PMID 20045849